CLINICAL TRIAL: NCT00921674
Title: A Single-dose, Randomised, Crossover Study to Compare the Rate and Extent of Absorption of Two Formulations of Ivermectin in Healthy Male and Female Volunteers After Food
Brief Title: Ivermectin Solution Bioequivalence Study - With Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SCO2804
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: therapeutic equivalency; pharmacokinetics; food; Healthy Volunteers
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ivermectin (Experimental): ivermectin
  Interventions: Drug: ivermectin

INTERVENTIONS:
Drug: ivermectin — Each subject will receive single doses of (i) 30 ml ivermectin oral solution (30 mg) and (ii) 10 x 3 mg tablets of ivermectin (30 mg) in 2 separate dosing periods. Doses will be administered 20 minutes after a standard breakfast.
  Other Names: Stromectol

SUMMARY:
The purpose of this study was to compare the pharmacokinetic and bioavailability profile (rate and amount of absorption into the bloodstream) of a test formulation of Ivermectin solution 1 mg/ml with a marketed reference formulation of Ivermectin 3 mg tablets when taken after a standard meal. The study is designed in accordance with the EU Note for Guidance on the Investigation of Bioavailability and Bioequivalence 2001.

DETAILED DESCRIPTION:
Ivermectin is an antiparasitic medicine (i.e. a medicine used to eliminate parasitic worms) for oral administration, and is approved in the US and some other countries in a tablet form. A new liquid formulation of ivermectin has been developed to facilitate dosing. This is a single dose, randomised, crossover study in healthy adult male and female volunteers, with doses taken 20 minutes after a standard breakfast. Doses will be separated by washout period of at least 14 days. Twenty-one blood samples will be taken from each volunteer over 144 hours in each period. Concentrations of Ivermectin in plasma will be measured using a validated chromatographic assay (LC-MS/MS). Standard pharmacokinetic parameters will be obtained and bioequivalence on the basis of rate and extent of drug absorption will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Aged between 18 and 50 years
* BMI </= 30 kg/m2
* Weight between 50 and 90 kg
* Non-smokers, or smokers of fewer than 10 cigarettes per day
* Clinically normal medical history
* Clinically normal findings on physical examination
* Clinically normal blood pressure ( >/= 100/60 for males; >/= 90/50 for females; </= 140/90 for both)
* Electrocardiogram recording (12-lead) within the normal range
* Clinically normal findings for haematology and clinical chemistry of blood and urine, or showing clinically insignificant deviations only
* Negative screening results (within the 14 days before study start) for drug of abuse, including opiates, cannabinoids, amphetamines, methamphetamine, benzodiazepines and cocaine
* Negative HIV and Hepatitis B and C tests (within the 14 days before study start)
* Appropriate use of an effective method of contraception (female volunteers only)
* Negative pregnancy test (female volunteers only)
* Ability to comprehend and communicate effectively with the Investigator and staff
* Ability to give written informed consent

Exclusion Criteria:

* Illness within 14 days before the start of the study
* Hospitalisation within 3 months before the start of the study (at the discretion of the Investigator)
* Participation in a clinical trial in which blood was taken within 16 weeks before the start of the study
* Participation in a clinical trial in which a volume of blood exceeding 500 ml was taken within 12 months before the start of the study
* Donation of blood or plasma within 90 days before the start of the study
* Any indication of current or previous abuse of alcohol, solvents or drugs
* Treatment with a full or regular course of medication during the 28 days before the start of the study or with any proscribed medication during the 14 days before the start of the study
* Use of alcohol on study days or within 24 hours prior to commencement of each study period
* Intake of grapefruit products within 7 days before the start of the study
* Intake of methylxanthine-containing beverages within 24 hours prior to each study period
* Intake of quantities of methylxanthine or alcohol-containing beverages which, in the opinion of the Investigator are abnormal (habitually taking more than 5 cups or glasses of tea, coffee, cola, chocolate etc. per day or habitually taking more than 20 g alcohol/day)
* Patient is pregnant, or lactating/breastfeeding (female volunteers only)
* Diet, which in the opinion of the Investigator, deviates from a normal diet (e.g. vegans)
* Patients who have resided in areas of Africa known to be endemic for Onchocerca volvulus (onchocerciasis or river blindness), wuchereria bancrofti (lymphatic filariasis), Loa loa or other microfilaremic disease
* Patients with a known or suspected intestinal helminth infection, such as Strongyloides stercoralis or other intestinal helminth
* Patients with a known hypersensitivity to any component of the Ivermectin product

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, including AUC0-t, AUC0-inf, and Cmax | 21 samples over 144 hours in each period, with a 14-day washout

SECONDARY OUTCOMES:
Pharmacokinetic parameters, including t1/2, Mean residence time (MRT), Terminal Elimination Rate Constant (kel) and Tmax | 21 samples over 144 hours in each period, with a 14-day washout

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Cottrell, Study Director — McNeil UK